CLINICAL TRIAL: NCT00565396
Title: Multi-Center,Double-Blind,Randomized,Controlled Clinical Trial of Fosinopril and/or Losartan in Patients With Chronic Kidney Disease Stage 3
Brief Title: Effectiveness Study on Fosinopril and/or Losartan in Patients With Chronic Kidney Disease Stage 3
Acronym: FLIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Municipal Health Bureau (Other Government)
Responsible Party: Nan Chen, Ruijin Hospital, Shanghai Jiao Tong University, School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2003ZD002; 2003ZD002
Record Dates: First submitted 2007-11-28; First posted 2007-11-30 (Estimated); Last update posted 2007-11-30 (Estimated); Status verified 2007-11

CONDITIONS: Chronic Kidney Insufficiency; Angiotensin-Converting Enzyme Inhibitors; Angiotensin II Type 1 Receptor Blockers; Proteinuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — Fosinopril; Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Fosinopril 10mg/day(oral)
  Interventions: Drug: Fosinopril and Losartan
- 2 (Active Comparator): Fosinopril 20mg/day(oral)
  Interventions: Drug: Fosinopril and Losartan
- 3 (Active Comparator): Losartan 50mg/day(oral)
  Interventions: Drug: Fosinopril and Losartan
- 4 (Active Comparator): Losartan 100mg/day(oral)
  Interventions: Drug: Fosinopril and Losartan

INTERVENTIONS:
Drug: Fosinopril and Losartan — Fosinopril 10mg/day(oral) Losartan 50mg/day(oral)

SUMMARY:
The purpose of this study is to determine whether fosinopril and losartan are effective in the treatment of patients with Chronic Kidney Disease(CKD) stage 3.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years old
* Roll out secondary renal diseases
* Do not use steroids and immunosuppresive drugs
* ACEI/ARB treated patients should have 7-14 days wash out period，SiDBP< 110mmHg
* Willing and able to comprehend and give written informed consent
* Willing to follow-up regularly

Exclusion Criteria:

* Use steroids and immunosuppresive drugs
* Secondary renal diseases
* Acute cardio-cerebral diseases within 6 months
* Post renal transplantation
* Pregnant/Nursing women
* History of hypersensitivity to ACEI/ARB
* Refuse to join clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2004-09; Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
progress to End Stage Renal Disease | within two years
double of serum creatinine | within two years
all cause mortality | within two years

SECONDARY OUTCOMES:
decreased proteinuria | within two years

CONTACTS AND LOCATIONS:
Overall Officials: Nan Chen, M.D., Study Chair — Ruijin Hospital
Locations (26):
- China (26):
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - The 1st Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Guangxing Hospital, Hangzhou, Zhejiang
  - Shaoyifu Hospital, Hangzhou, Zhejiang
  - Ningbo Lihuili Hospital, Ningbo, Zhejiang
  - Wenling 1st People's Hospital, Wenling, Zhejiang
  - The First affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang
  - Xiangshan People's Hospital, Xiangshan, Zhejiang
  - Renji Hospital, Shanghai
  - Changzheng Hospital, Shanghai
  - Shanghai 9th People's Hospital, Shanghai
  - Ruijin Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai
  - Zhongshan Hospital, Shanghai
  - Huadong Hospital, Shanghai
  - Huashan, Shanghai
  - Shanghai 455 Hospital, Shanghai
  - Shanghai 85 Hospital, Shanghai
  - Tongji Hospital, Shanghai
  - Shanghai 10th People's Hospital, Shanghai
  - Shanghai 1st People's Hospital, Shanghai
  - Shanghai Yangpu District Centre Hospital, Shanghai
  - Xinhua Hospital, Shanghai
  - Shanghai East Hospital, Shanghai
  - Shanghai 6th people's hospital, Shanghai
  - Shanghai Changning District Centre Hospital, Shanghai
  - Changhai Hospital, Shanghai